CLINICAL TRIAL: NCT05776615
Title: The Effect of the Mobile Application Developed for the Care of Sick Newborns on Nurses' Perception of Nursing Diagnoses and MissCare: A Randomized Controlled Trial
Brief Title: The Effect of the Mobile Application Developed for the Care of Sick Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: HF-22003
Record Dates: First submitted 2023-02-15; First posted 2023-03-20 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Nursing Caries; Newborn
Keywords: Newborn; Misscare; Nursing Process; Mobile Application

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental study
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application Group (Experimental): In the collection of Mobile Application data, they will be asked to fill out the forms.The mobile application will be introduced, the application will be downloaded from the virtual market (Google Play Store or App Store) to the phone, login will be provided by giving a user name and password, and how to use the application will be explained. Participants will be asked to provide nursing care using this application once a week for 3 months. Nursing Diagnosis Perception Scale with nurses at the end of the 1st month and at the end of the 3rd month; " MıssCare" Detection Questionnaire in the Neonatal Intensive Care Unit; System Availability Scale will be applied.
  Interventions: Other: mobile application
- Control group (No Intervention): Participants included in the control group, Nurse Descriptive Characteristics form; Nursing Diagnoses Perception Scale, "Missing Nursing Care" Detection Questionnaire will be applied in the Neonatal Intensive Care Unit. Nursing Diagnoses Perception Scale at the end of the 1st month and at the end of the 3rd month; The "Missing Nursing Care" Identification Questionnaire will be applied again in the Neonatal Intensive Care Unit, and the System Usability Scale will not be applied to the control group.

INTERVENTIONS:
Other: mobile application — In the collection of Mobile Application group data, they will be asked to fill out the forms.The mobile application will be introduced, the application will be downloaded from the virtual market (Google Play Store or App Store) to the phone, login will be provided by giving a user name and password, and how to use the application will be explained. Participants will be asked to provide nursing care using this application once a week for 3 months.Nursing Diagnosis Perception Scale with nurses at the end of the 1st month and at the end of the 3rd month; " MıssCare" Questionnaire in the Neonatal Intensive Care Unit(NICU); System Availability Scale will be applied.
  Arms: Mobile Application Group

SUMMARY:
The goal of this randomize controlled trial determine the effect of the mobile application developed for the care of sick newborns in the Neonatal Intensive Care Unit on nurses' perception of nursing diagnoses and care that cannot be met, and to measure the usability of the mobile application. The main questions it aims to answer are; Does the mobile application developed for the care provided in the neonatal intensive care unit have an effect on the perception of nursing diagnoses? Does the mobile application developed for care provided in the neonatal intensive care unit have an impact on "missed nursing care? Participants will be used for 3 months from the developed mobile application. The control group will continue routine nursing care.

Researchers will compare the perception of nursing diagnosis and unaffordable nursing care survey at the end of month 1 and month 3. Additionally, the usability of the mobile application will be evaluated by applying the system applicability scale to the experimental group.

DETAILED DESCRIPTION:
Mobile application has become an important and necessary element in nursing education and clinical nursing practices, and its use has gradually increased. Neonatal intensive care units (NICUs) are areas where complex and quality health care is provided for newborns. The development of the nursing process, especially in the neonatal intensive care unit, may shorten the duration of the care that should be provided to newborns. New ways such as mobile applications can be sought to assist in the realization of the nursing process and to strengthen the diagnostic perception of neonatal nurses. This study is a randomized controlled experimental study designed to determine the effect of the mobile application developed for the care of sick newborns in the Neonatal Intensive Care Unit on nurses' perception of nursing diagnoses and care that cannot be met, and to measure the usability of the mobile application. A total of 69 nurses working in the neonatal intensive care unit in turkey will constitute the universe of the research. In this study, participants will be selected for experimental and control groups using a stratified random sampling method (the stratification criteria will be based on the institutions where the nurses work). The sample will be calculated as experimental group: 27 control group: 27 in total. Samples from the identified will be selected using the random numbers table.

In this study, Nurse Descriptive Characteristics Form; Nursing Diagnosis Perception Scale ; Questionnaire for Determining "missed nursing care" in the Neonatal Intensive Care Unit created by the researcher ; System Usability Scale will be used. For the missed nursing care nursing care determination questionnaire, expert opinion was taken and applied to the pilot group, and its content validity was checked.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working actively in NICU,
* Active user nurses who have a smart phone with IOS or Android software.

Exclusion Criteria:

* Failed to complete all the steps of the research,
* Nurses who want to leave the research voluntarily

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seher SARIKAYA KARABUDAK, Ass.Prof., Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University, Aydin, EFELER, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almeida SR, Sasso GT, Barra DC. Computerized nursing process in the Intensive Care Unit: ergonomics and usability. Rev Esc Enferm USP. 2016 Nov-Dec;50(6):998-1004. doi: 10.1590/S0080-623420160000700017. English, Portuguese. PMID 28198966
- [Background] Amoakoh-Coleman M, Borgstein AB, Sondaal SF, Grobbee DE, Miltenburg AS, Verwijs M, Ansah EK, Browne JL, Klipstein-Grobusch K. Effectiveness of mHealth Interventions Targeting Health Care Workers to Improve Pregnancy Outcomes in Low- and Middle-Income Countries: A Systematic Review. J Med Internet Res. 2016 Aug 19;18(8):e226. doi: 10.2196/jmir.5533. PMID 27543152
- [Background] Asif M, Jameel A, Hussain A, Hwang J, Sahito N. Linking Transformational Leadership with Nurse-Assessed Adverse Patient Outcomes and the Quality of Care: Assessing the Role of Job Satisfaction and Structural Empowerment. Int J Environ Res Public Health. 2019 Jul 4;16(13):2381. doi: 10.3390/ijerph16132381. PMID 31277478
- [Background] Baccin CRA, Dal Sasso GTM, Paixao CA, de Sousa PAF. Mobile Application as a Learning Aid for Nurses and Nursing Students to Identify and Care for Stroke Patients: Pretest and Posttest Results. Comput Inform Nurs. 2020 Jul;38(7):358-366. doi: 10.1097/CIN.0000000000000623. PMID 32427611
- [Background] Basch E, Artz D, Iasonos A, Speakman J, Shannon K, Lin K, Pun C, Yong H, Fearn P, Barz A, Scher HI, McCabe M, Schrag D. Evaluation of an online platform for cancer patient self-reporting of chemotherapy toxicities. J Am Med Inform Assoc. 2007 May-Jun;14(3):264-8. doi: 10.1197/jamia.M2177. Epub 2007 Feb 28. PMID 17329732
- [Background] Bautista JR. Filipino Nurses' Use of Smartphones in Clinical Settings. Comput Inform Nurs. 2019 Feb;37(2):80-89. doi: 10.1097/CIN.0000000000000482. PMID 30299305
- [Background] Bautista JR, Lin TT. Sociotechnical analysis of nurses' use of personal mobile phones at work. Int J Med Inform. 2016 Nov;95:71-80. doi: 10.1016/j.ijmedinf.2016.09.002. Epub 2016 Sep 16. PMID 27697234
- [Background] Bhatheja S, Fuster V, Chamaria S, Kakkar S, Zlatopolsky R, Rogers J, Otobo E, Atreja A, Sharma SK, Kini AS. Developing a Mobile Application for Global Cardiovascular Education. J Am Coll Cardiol. 2018 Nov 13;72(20):2518-2527. doi: 10.1016/j.jacc.2018.08.2183. PMID 30442294
- [Background] Blackman I, Henderson J, Willis E, Hamilton P, Toffoli L, Verrall C, Abery E, Harvey C. Factors influencing why nursing care is missed. J Clin Nurs. 2015 Jan;24(1-2):47-56. doi: 10.1111/jocn.12688. Epub 2014 Sep 30. PMID 25265893
- [Background] Blackman I, Lye CY, Darmawan IGN, Henderson J, Giles T, Willis E, Toffoli L, Xiao L, Verrall C. Modeling Missed Care: Implications for Evidence-Based Practice. Worldviews Evid Based Nurs. 2018 Jun;15(3):178-188. doi: 10.1111/wvn.12285. Epub 2018 Mar 23. PMID 29569380
- [Background] Blackman I, Papastavrou E, Palese A, Vryonides S, Henderson J, Willis E. Predicting variations to missed nursing care: A three-nation comparison. J Nurs Manag. 2018 Jan;26(1):33-41. doi: 10.1111/jonm.12514. Epub 2017 Jul 27. PMID 28752529

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Inclusion Criteria for the Study:Nurses' inclusion criteria for the study; Nurses who were actively working in the NICU, had an IOS or Android smartphone, and were active users were included in the study.
  Exclusion Criteria for the Study:Nurses who had a Windows or Blackberry smartphone were not included in the study.
  Exclusion Criteria for the Study:Nurses who could not complete all the steps of the study and who wanted to leave the study of their own volition were excluded from the study.
Period: Overall Study
Arm/Group | Mobile Application Group | Control Group
Started | 32 | 32
Completed | 31 | 32
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Newborn nurse
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Application Group | Control Group | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 32 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 31 | 32 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 31 | 32 | 63
Region of Enrollment [Number; unit: participants]
  Turkey | 31 | 32 | 63
Professional working time [Count of Participants; unit: Participants] — Less than 1 year 1-5 years More than 5 years
  Participants
    Less than 1 year | 1 | 2 | 3
    1-5 years | 7 | 4 | 11
    More than 5 years | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Pre-test The Nurse Descriptive Characteristics Form; The Nursing Diagnoses Perception Scale; MissCare Nursing Care Questionnaire in the Neonatal Intensive Care Unit
Description: Nurse Descriptive Characteristics Form: A 19-item questionnaire (18 closed, 1 open-ended) developed from the literature to collect demographic and professional information including education, experience, NICU background, work schedule, caregiving practices, nursing process use, and mobile app use. Scoring: Descriptive only.
  Nursing Diagnosis Perception Scale: A 20-item, 5-point Likert scale (1 = Strongly agree, 5 = Strongly disagree) assessing four subscales-Professional definition, Clarity, Ease of use, Conceptual dimension. Score range: 1-5 (mean). Lower scores indicate more positive perceptions.
  MissCare Nursing Care Questionnaire in the NICU: A 69-item, 4-point Likert tool (1 = Always performed, 4 = Never performed) evaluating missed care in ten domains; lower scores reflect more complete care.
Time Frame: Before starting the intervention
Population: 1 person left her job due to pregnancy
Measure: Median (Standard Deviation); unit: units on a scale
Groups:
- Mobile Application Group; Control Group: In the study, before the mobile application , the overall score of the study group was 2.44±0.28, while the control group was 2.44±0.29.
Arm/Group | Mobile Application Group | Control Group
Number analyzed (Participants) | 31 | 32
units on a scale
  nursing diagnoses perception scale | 2.44 (0.28) | 2.44 (0.29)
  MissCare nursing care questionnaire | 1.16 (0.18) | 1.12 (0.14)

2. Primary Outcome: 1. The Nursing Diagnoses Perception Scale 2. MissCare Nursing Care Questionnaire in the Neonatal Intensive Care Unit 3. System Usability Scale-Turkish (SUS-TR)
Description: Nursing Diagnosis Perception Scale: A 20-item, 5-point Likert scale (1 = Strongly agree, 5 = Strongly disagree) assessing four subscales-Professional definition, Clarity, Ease of use, Conceptual dimension. Score range: 1-5 (mean). Lower scores indicate more positive perceptions.
  MissCare Nursing Care Questionnaire in the NICU: A 69-item, 4-point Likert tool (1 = Always performed, 4 = Never performed) evaluating missed care in ten domains; lower scores reflect more complete care.
  System Usability Scale-Turkish (SUS-TR) is a brief scale developed to measure user views on system usability. Scores are calculated on a 0-100 scale, with higher scores indicating better usability. "This scale was applied exclusively to the Mobile Application Group.
Time Frame: 1 Months
Population: In the 1st month she stopped working due to pregnancy.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Application Group | Control Group
Number analyzed (Participants) | 31 | 32
units on a scale
  MissCare nursing care questionnaire | 1.14 (0.14) | 1.14 (0.15)
  nursing diagnoses perception scale | 2.31 (0.42) | 2.36 (0.33)
  System Usability Scale | 86.90 (12.63) | 0 (0)

3. Secondary Outcome: 1. The Nursing Diagnoses Perception Scale 2. MissCare Nursing Care Questionnaire in the Neonatal Intensive Care Unit 3. System Usability Scale-Turkish (SUS-TR)
Description: as for outcome 2
Time Frame: 3 months
Population: no casualties
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Group; Mobile Application Group: Before using the mobile app, the study and control groups had similar HTAQ general scores , with no significant difference (p>0.05). However, the study group showed significant changes over time ), with lower scores at the 1st and 3rd months compared to the pre-test. No significant changes were observed in the control group. Both groups showed no significant difference in NICU NICU NICU scores (p>0.05). In the study group, NICU HRBA scores significantly decreased over time, with the 1st month and pre-test scores higher than the 3rd month. The control group also showed a significant difference in NICU HRQL scores, but no change between the 1st and 3rd month scores. In the NICU, the 1st-month scores were significantly higher than the 3rd-month scores.
Arm/Group | Control Group | Mobile Application Group
Number analyzed (Participants) | 32 | 31
units on a scale
  Nursing Diagnoses Perception Scale:Diagnoses Perception Scale | 2.25 (0.42) | 2.19 (0.29)
  NICU MissCare Nursing Care Questionnaire | 1.10 (01.2) | 1.07 (0.12)
  System Usability Scale-Turkish (SUS-TR) | 0 (0) | 86.13 (13.18)

ADVERSE EVENTS:
Time Frame: 3 month
Arm/Group | Mobile Application Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

LIMITATIONS AND CAVEATS:
This study included nurses with smartphones running Android or iOS. The collection of personal information (name and surname) may have influenced their responses, and nurses might have provided biased answers due to concerns about their image with managers. Additionally, the simultaneous presence of both study and control group nurses in the clinic may have led to information sharing between the groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/15/NCT05776615/Prot_SAP_ICF_000.pdf